CLINICAL TRIAL: NCT07107581
Title: A Post-Market Domestic (US) and International Data Collection to Assess Exactech Knee Systems
Brief Title: Exactech Knee Systems Post Market Clinical Follow-up
Status: Enrolling by invitation | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: TM- 2022-012696
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Knee Arthroplasty, Total; Partial Knee Replacement
Keywords: Exactech; Knee Arthroplasty
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Cohort 1. Prospective / Subjects Knee Arthroplasty: Enrolled in the study pre-surgery
  Interventions: Device: Prospective / Subjects Knee Arthroplasty
- Cohort 2. Retrospective to Prospective: Subjects enrolled in the study post- surgery then continue to participate in the study prospectively.
  Interventions: Device: Retrospective to Prospective
- Cohort 3. Retrospective Only Subjects: Enrolled in the study post-study surgery with no intent to continue as prospective subjects.
  Interventions: Device: Retrospective Only Subjects

INTERVENTIONS:
Device: Prospective / Subjects Knee Arthroplasty — Knee Arthroplasty
  Groups: Cohort 1. Prospective / Subjects Knee Arthroplasty
Device: Retrospective to Prospective — Knee Arthroplasty
  Groups: Cohort 2. Retrospective to Prospective
Device: Retrospective Only Subjects — Knee Arthroplasty
  Groups: Cohort 3. Retrospective Only Subjects

SUMMARY:
This is a multi-center, open-label, prospective and retrospective clinical outcomes study. Patient outcomes data is important for assessing the post-market safety and effectiveness of orthopedic medical devices. The purpose of this study is to collect clinical and patient outcomes and survivorship data for patients who have received or will receive an Exactech Knee System total knee arthroplasty (TKA) prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA).

Subjects will, or will have already, undergo/undergone TKA as prescribed by the operating surgeon in a medical center with appropriate facilities and appropriately trained personnel. Treatment will be with the knee replacement components described in this protocol. The surgical procedure shall be conducted according to the appropriate Surgical Technique (Reference #: 712-35-41 and 712-35-35 as applicable) and product labeling for an Exactech Knee System and in accordance with the standard of care of the operating surgeon.

The medical devices and procedures used in this study are considered standard of care and are not considered investigational or experimental.

Information about the subject's preoperative conditions, demographics, previous surgical procedures, devices used, surgical procedure, postoperative outcomes, radiographic outcomes, and adverse events should be collected according to the Protocol Activity Schedule below:

Cohort 1. Prospective Subjects Enrolled in the study pre-surgery:

Cohort 2. Retrospective-to-Prospective Subjects - Subjects Enrolled in the study post-surgery.

Cohort 3. Retrospective Only Subjects - Data collection for the Retrospective Only Subjects will occur through a retrospective, observational, medical chart review.

Visit & Windows of data to be collected for all Cohorts:

* Preoperative Visit- Within ≤ 3 months prior to surgery
* Surgery/Discharge -Day of Surgery /Day of Discharge
* 6 Week Post-Op Visit - (Porous cohort only) -3 weeks - 7 weeks
* 6 Month Post-Op Visit - (Required for porous, optional for cemented) - 8 weeks - 26 weeks
* 1 through 10 Year Post-Operative Follow-Up Visits (As per the surgeon's standard of care) - ±6 months

Clinical Outcomes to be collected (only if available for Cohort 3):

* Functional Performance
* Range of Motion

  1. Patient Outcomes to be collected (only if available for Cohort 3):
* Knee injury and Osteoarthritis Outcome Score for Joint Replacement Jr. (KOOS Jr.)
* Knee Society Score (KSS) / Hospital for Special Surgery Score (HSS)
* Oxford Knee Score (OKS)
* Visual Analog Scale (VAS) for Pain and Patient Satisfaction

  2. Safety Outcomes:

  a. Adverse Events
* Procedure-related adverse events,
* Device related adverse events,
* Readmissions, and Revisions b. Radiographic Outcomes (Assessment) (e.g., radiolucent lines, subsidence) c. Survivorship Rates - Kaplan Meier Analysis with a survivorship distribution function

DETAILED DESCRIPTION:
3. Sample Size and Justification

Enrollment targets are based on, but not limited to, a sample size of 1879 primary subjects. Subjects will be enrolled based on a statistical estimation of the sample size needed to examine the primary outcome of survivorship (i.e., implant revision). The below table describes the distribution of enrollment. Additional subjects and component types may be enrolled beyond those described below.

1. Truliant CR, n=308 Cemented Femoral, n=154 Porous Femoral, n=154 Tibial Insert CR, n=154 Tibial Insert CRC, n=154
2. Truliant PS, n=610 Cemented Femoral, n=305 Porous Femoral, n=305 Tibial Insert PS, n=305 Tibial Insert PSC, n=305
3. Logic CR, n=308 Cemented Femoral, n=154 Porous Femoral, n=154 Tibial Insert CR, n=154 Tibial Insert CRC, n=154
4. Logic PS, n=610 Cemented Femoral, n=305 Porous Femoral, n=305 Tibial Insert PS, n=305 Tibial Insert PSC, n=305
5. Constrained Condylar Components, n=43 CC Cemented Femoral Components, n=43 CC Tibial Inserts, n=43

   Each product's subgroups share the same parameters and assumptions resulting in equal sample size. Sample sizes are estimated by component to ensure sufficient clinical data on each Total Knee Arthroplasty (TKA) component from each system. Because a patient must undergo a TKA with both a tibial insert and a femoral component, that individual patient will count toward the sample size for each component. All calculations consider an estimated 40% attrition rate.

   The sample size calculations indicate the estimated width of the 95% confidence limits for the primary endpoint, namely implant survivorship at 10 years, based on data obtained from the literature. The calculation generated a proposed sample size sufficient to support a 10-year survivorship analysis. To ensure data consistency and quality across the planned study time points, the sample size estimation is applied to the prospectively enrolled subjects only.

   4. Data Collection

   Standard follow-up visits should be conducted to collect ongoing subject outcomes data. Electronic Patient Reported Outcomes (ePRO) may be available for subjects/sites to use for collection of safety data and patient reported outcomes.

   5. Data Collection Forms/Logs

   Paper Case Report Forms (CRFs) will be provided to assist sites with data collection, if requested. The use of paper CRFs may be implemented into the site's workflow completely, partially, or not at all. All data submitted to Exactech through an eCRF within the EDC must be verifiable in the patient's medical records or paper CRF. The original source of data submitted via electronic case report forms (eCRFs) for this study must be established prior to data collection.

   6. Data Recording:

   An electronic data capture (EDC) system will be used for recording data in this study. The EDC system provides an electronic version of the paper forms that allow for simple online completion and submission of the forms. The EDC system can be accessed from any computer with internet capabilities and provides a secure internet connection for data entry.

   Each site will need to be assigned login information (User ID and Password) from Exactech to access the forms. Sites will also be provided with the paper forms, if requested, so that all appropriate data can be collected during each subject visit. The data collected on the paper forms can then be used to complete the online (Internet) forms.

   7. Data Quality Assurance

   Investigative sites will be notified of incomplete or discrepant data so that corrections or additional data can be provided, as appropriate. Whether a site is using paper or electronic forms it is important to fill out each form as completely, legibly, and accurately as possible before submitting it to the Sponsor via eCRF.

   8. Outcome Assessment

   Analysis of clinical outcomes will be summarized using appropriate descriptive statistics (means, standard deviations, medians, minimum and maximums for continuous variables, and percentages for categorical variables at each point in time).

   9. Device Survival

   A Kaplan-Meier survival curve analysis will be performed to account for variability in length of follow- up.

   10. Complications

   Device-related complications, both "possibly," and "definitely" related, as well as serious adverse events will be summarized by reporting the total number of reported events by the number of operative cases.

   11. Study Monitoring

   Study monitoring will occur according to the Monitoring Plan set out specific to this study. The monitoring duties are to aid the Clinical Investigator in the production and maintenance of complete, legible, well-organized, and easily retrievable data. In addition, the Monitor will be responsible for ensuring the Clinical Investigators' understanding of the CIP and all applicable regulations.

   12. Good Clinical Practices (GCP)

   This investigation will be conducted in accordance with the principles of BS EN International Organization for Standardization (ISO) 14155:2020 titled "Clinical investigation of medical devices for human subjects" and International Council for Harmonisation (ICH) GCP (Good Clinical Practice) guidelines.

ELIGIBILITY:
Cohort 1. Prospective / Subjects

Enrolled in the study pre-surgery:

Subjects who agree to participate in the study have not had surgery prior to being enrolled in the study.

Skeletally mature (18 years of age or older).

The subject is willing and able to provide written informed consent for participation in the study.

Subject is to receive an Exactech Knee System TKA for any approved indication for use.

The knee replacement will be performed by the investigator or a sub- investigator.

The devices will be used according to the approved indications.

Cohort 2. Retrospective to Prospective

Subjects enrolled in the study post- surgery then continue to participate in the study prospectively.

Subjects who agree to participate, who have had surgery prior to enrollment in the study. Data for these subjects will be collected from the subject's medical record for the time-period prior to enrollment in the study containing data pertaining to the preoperative time period and index surgery (retrospective data) and from the patient after they are enrolled in the study during the post-operative time-period (prospectively).

Skeletally mature (18 years of age or older).

The subject is willing and able to provide written informed consent for participation in the study.

Subject received an Exactech Knee System TKA for any approved indication for use.

The knee replacement was performed by the investigator or a surgeon sub-investigator.

The devices are/were used according to the approved indications.

Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria, and have a minimum of the following pre- operative, operative, and applicable postoperative data available in the subject's medical records, related to the Exactech Knee System prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for data submission:

Pre-Operative:

Demographic Data

Gender

Age at surgery

Height/Weight

Indication for surgery

Prior Injuries/Surgeries on index knee

Comorbidities

Operative:

Date of Surgery

Type of Surgery (Primary / Revision)

All component product information, including catalogue reference numbers.

Adverse Event Information, if applicable

Cohort 3. Retrospective Only Subjects

Enrolled in the study post-study surgery with no intent to continue as prospective subjects.

Note: No prospective data may be collected from a subject if they are enrolled under this cohort unless the subject is willing and able to provide written informed consent for participation in the study, in which case they should be part of Cohort 2.

Skeletally mature at the time of the surgery (18 years of age or older).

The patient's clinical record includes a signed waiver that clearly expresses patient consent for the use of available clinical data for the purpose of clinical research outside of the operating institution.

The patient's clinical record includes a documented procedure that includes, or is related to, TKA with an Exactech Knee System device.

The knee replacement was performed by the investigator or a surgeon sub-investigator.

The devices are/were used according to the approved indications.

Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria and have a minimum of the following pre- operative, operative, and applicable postoperative data available in the subject's medical records, related to the Exactech Knee System prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for submission:

Pre-Operative:

Demographic Data

Gender

Age at surgery

Height/Weight

Indication for surgery

Prior Injuries/Surgeries on index knee

Comorbidities

Operative:

Date of Surgery

Type of Surgery (Primary / Revision)

All component product information, including catalogue reference numbers.

Adverse Event Information, if applicable

Exclusion Criteria:

Patient was <18 years of age at time of surgery Patient does not meet indicated population for use criteria for this device. Patient is pregnant Patient is a prisoner Patient has a physical or mental condition that would invalidate the results Patient is contraindicated for the surgery (e.g., metal allergy)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject received or is to receive an Exactech Knee System TKA for any approved indication for use.
Sampling Method: Probability Sample
Enrollment: 1879 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 10 Years
  The objective of this study is to assess the safety and performance of Exactech Knee System devices. Data will be collected to provide objective evidence of safety and performance of Exactech Knee Systems used in primary knee arthroplasty. Data may be analyzed to support future presentations and publications of an Exactech Knee System and may be used to provide clinical evidence of the post market outcomes of Exactech Knee Systems to regulatory authorities when required.
  The following data will be collected:
  Demographics (e.g., height, weight, age, and gender), Preoperative information (e.g., indication for surgery, comorbidities, pre-surgical assessments of knee function), Operative details (e.g., intra-operative findings, surgical approach, length of surgery), Product information (components used in the knee surgery), Adverse events (e.g., infection, device failure, revision), Implant survivorship, & Patient Reported Outcomes (KOOS, KSS, HSS, OKS and/or VAS)

SECONDARY OUTCOMES:
Secondary Objective | 10 Years
  Collect radiographic data when available to examine radiographic outcomes. Analyze safety and performance of Exactech Knee System components when used in revision cases. Appropriate radiographs should be obtained to allow proper evaluation of the knee(s) by the investigator. The evaluation of the radiographs should be documented on the appropriate case report form for each applicable visit.
  1. Radiographic views include:
     1. AP View (weight bearing)
     2. Lateral View
     3. Patellar Skyline or Merchant View
  2. Radiographic evaluations include:
     1. Preoperative visit
     2. Immediate postoperative visit
     3. Post-operative follow-up visits
  3. Radiographic assessments include:
     1. Knee alignment
     2. Patellofemoral evaluation
     3. Radiolucent lines
     4. Subsidence

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Rohrs, PhD, Study Director — Exactech
Locations (1):
- Florida Orthopaedic Associates, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns related to patient privacy, data confidentiality, and regulatory restrictions. Additionally, data sharing agreements or consent obtained from participants may not permit the broad dissemination of IPD

REFERENCES:
- [Background] Martin A, Quah C, Syme G, Lammin K, Segaren N, Pickering S. Long term survivorship following Scorpio Total Knee Replacement. Knee. 2015 Jun;22(3):192-6. doi: 10.1016/j.knee.2015.01.007. Epub 2015 Mar 26. PMID 25818502
- [Background] Scott CE, Clement ND, MacDonald DJ, Hamilton DF, Gaston P, Howie CR, Burnett R. Five-year survivorship and patient-reported outcome of the Triathlon single-radius total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1676-83. doi: 10.1007/s00167-014-2922-8. Epub 2014 Mar 13. PMID 24623184
- [Background] Meftah M, White PB, Ranawat AS, Ranawat CS. Long-term results of total knee arthroplasty in young and active patients with posterior stabilized design. Knee. 2016 Mar;23(2):318-21. doi: 10.1016/j.knee.2015.10.008. Epub 2016 Jan 29. PMID 26833096